CLINICAL TRIAL: NCT06131541
Title: Alveolar Ridge Splitting With Simultaneous Implant Placement Using Undemineralized Autogenous Tooth Graft: a Randomized Clinical Trial
Brief Title: Ridge Splitting With Implant Placement Using Autogenous Tooth Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Assistant Professor of periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-80
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Dental Implant Failure Nos; Alveolar Bone Loss; Peri-Implantitis
Keywords: Ridge splitting; Autogenous Tooth Graft; simultaneous implant placement
MeSH Terms: conditions — Alveolar Bone Loss; Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: single-center, prospective, single-blinded, randomized parallel two-arm controlled clinical trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The present clinical trial was single-blinded one as the evaluator and the statistician were both blinded. While both the implantologist or the participant were not blinded as the interventions were dissimilar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: autogenous bone graft group (Experimental): 11 subjects will be assigned to receive alveolar ridge splitting in combination with autogenous bone graft associated with immediate implant placement
  Interventions: Procedure: autogenous bone graft
- Group II: autogenous tooth graft group (Experimental): 11 subjects will be assigned to receive alveolar ridge splitting in combination with undemineralized autogenous tooth graft associated with immediate implant placement
  Interventions: Procedure: autogenous tooth graft

INTERVENTIONS:
Procedure: autogenous tooth graft — undemineralized autogenous tooth graft will augment the gap between the splitted ridge and the simultaneously [laced implant fixture
  Arms: Group II: autogenous tooth graft group
Procedure: autogenous bone graft — autogenous bone graft will augment the gap between the splitted ridge and the simultaneously [laced implant fixture
  Arms: Group I: autogenous bone graft group

SUMMARY:
The aim of this study is to evaluate the radiographic and the clinical outcomes of application of the alveolar ridge splitting (ARS) in combination with ATG, associated with immediate implant placement versus ARS in combination with autogenous bone graft, associated with immediate implant placement in patients with horizontal bony insufficiency of alveolar ridges.

DETAILED DESCRIPTION:
In cases of a narrow ridge, the alveolar ridge expansion technique by means of hand osteotomes with gradually increasing dimensions was introduced by Tatum and modified by Summers and it can be used regardless of the bone quality.

Searching for absolute biocompatible material and taking into account the features of the enamel and dentin, using the tooth as an autologous grafting material was first advocated. Tooth and bone are sharing many characteristics, which supports the idea that tooth could be used as a grafting material. In fact, hydroxyapatite crystals make up the tooth inorganic composition (65%). Moreover, Collagen (mostly type I) and non-collagenic proteins comprised up the tooth organic component (35%). In addition, because autologous tooth graft (ATG) is denser than bone, minimal resorption rates were found to be advantageous to autobone. For the purpose of employing ATG as a grafting material, various methods and techniques have been suggested for developing undemineralized, demineralized or partially demineralized ATG.The outcomes of utilizing undemineralized autologous tooth graft (UATG) around SDIP following RSEA have not yet been evaluated. Therefore, the current trial aimed to assess the clinical and radiological performances of UATG for the treatment of horizontal alveolar ridge deficiencies using RSEA with SDIP.

The aim of this study is to evaluate the radiographic and the clinical outcomes of application of the alveolar ridge splitting (ARS) in combination with ATG, associated with immediate implant placement versus ARS in combination with autogenous bone graft, associated with immediate implant placement in patients with horizontal bony insufficiency of alveolar ridges.

ELIGIBILITY:
Inclusion Criteria:

* Good general health at the time of surgery
* At least 3 months of healing after tooth extraction
* Horizontally compromised alveolar ridges at least 10 mm high and 3 mm wide.

Exclusion Criteria:

* A vertical bone defect in the edentulous ridge;
* Thick cortex in the labial/buccal with less cancellous bone inside;
* Obvious undercut on the labial/buccal side;
* Uncontrolled periodontal conditions or other oral disorders;
* A history of radiotherapy in the head and neck region

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Stability Quotient of Implants (SQI) | 12-month.
  The implant stability was recorded using Osstell TM. Following implant insertion, SQI readings were taken immediately, then again after six and twelve months.
Horizontal bone dimensions (HBDs) | 12 months
  The HBD alterations were assessed by measuring horizontal spacing between the external edges of labial and palatal bony plates at a level 2mm apical of the fixture platform.
Peri-implant Bone Density (PBD) | 12 months
  For consistent measurement of the PBD, 1-mm-diameter Region of interest (RI) was selected and traced 1.2 mm distant from the fixture on the cross-sectional slices followed by counting the threshold pixels inside the RI.

SECONDARY OUTCOMES:
Pink esthetic score (PES) | 12 months
  Digital intraoral scannings were gathered before surgery, at 6 and 12-months after implantation, to evaluate the PES changes. Seven variables were assessed in relation to a nearby reference teeth: mesial and distal papilla, soft tissue level, colour, texture and shape, and alveolar bone defects. 14 is the maximum possible value for PES. Scoring each parameter on a 0-2 scale: 0 is the minimum score and 2 is the maximum.

CONTACTS AND LOCATIONS:
Overall Officials: WAlid AH Elamrousy, Ph.D, Principal Investigator — Kafrelsheikh University
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: No